CLINICAL TRIAL: NCT05253313
Title: Magnetic Resonance Imaging for Better Selection of Pancreatic Cancer Patients for Surgery
Brief Title: Magnetic Resonance Imaging for Better Selection of Pancreatic Cancer Patients for Surgery: A Randomized Clinical Trial
Acronym: MAGIPAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 22552255
Record Dates: First submitted 2022-02-01; First posted 2022-02-23 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-01

CONDITIONS: Pancreas Cancer
Keywords: Magnetic Resonance Imaging (MRi); Computed Tomography (CT)
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (No Intervention): Patients who are eligible for surgery are randomized to MRI scan or standard curative surgery. Patients in this arm will receive standard care according to danish standards without pre-operative MRI scans.
- MRI scan (Other): This arm includes patients who have been randomized to pre-operative MRI scans.
  Interventions: Other: MRI scan

INTERVENTIONS:
Other: MRI scan — Patients will be randomized to a pre-operative scan or not. The MRI scan will evaluate the local extent of the tumor and especially focus on identifying possible liver metastases unseen on the CT-scan.
  Arms: MRI scan

SUMMARY:
Pancreatic cancer has the most dismal prognosis with a 5-year survival of 8%. The only curative treatment is surgery which is accompanied by great morbidity and mortality. Recent research indicates that Magnetic Resonance Imaging (MRI) is superior in detecting liver metastases compared with today's gold standard computed tomography (CT), which usually is a contraindication to surgery.

Investigators want to randomize patients with pancreatic cancer, who are eligible for surgery to a pre-operative MRI. The investigators want to examine if MRI is as good for the staging as CT and if MRI is better for the identification of liver metastases. Patients will have a follow-up period of 1 year to see if MRI changes the overall survival.

DETAILED DESCRIPTION:
Currently, CT is the state of art for assessing and staging pancreatic cancer. However, it has its limitations when it comes to detecting small liver metastases, which are often found in pancreatic cancer. Recent research indicates that MRI is superior to CT when it comes to the detection of liver metastases. Thus, the investigators want to examine MRI's role in the assessment of pancreatic cancer.

The investigators want to conduct a nationwide RCT to examine the feasibility of using MRI for tumor staging and identification. The overall aim is to improve the selection of patients going to surgery so futile resections are avoided and increase the overall survival. Patients who are deemed eligible for pancreatic resection after being reviewed at a local multidisciplinary tumor board will be, upon consent, electronically randomized to one of two treatment arms (each arm will contain 100 patients). Patients within the control arm will as per usual proceed to surgery, whereas patients in the intervention arm will receive a pre-operative MRI scan. The MRI will be read by experienced gastroenterology radiologists who are blinded to the patient's identity and the initial CT findings. Treatment will be based on MRI findings. There will be a follow-up period of 1 year to see if MRI changes the overall survival. Within this RCT we will conduct three studies.

Study 1) The investigators want to compare pancreatic tumor staging with MRI versus standard upper abdominal CT, we hypothesize that MRI is not inferior to CT.

Study 2) The investigators want to assess MRI's ability to detect liver metastases vs standard upper abdominal CT, in patients otherwise deemed eligible for surgery. We hypothesize that MRI is superior to CT in the detection of liver metastases.

Study 3) The investigators want to assess the impact of MRI, thus patients will be followed for 1 year. We want to see if MRI changes the overall survival, treatment allocation, and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Must be eligible for curative pancreatic resection based on CT
* Must accept randomization

Exclusion Criteria:

* Not eligible for curative pancreatic resection
* Unable to undergo MRI.
* Did not accept randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Correlation in tumor staging (T- and N-stage) between CT and MR | 1 year
  The degree of correlation between CT and MR with respect to T- and N-stage. Will be assessed using Kappa-values.
Proportion of patients with liver metastases in the intervention arm | 1 year
  To examine if MRI scans identify more metastases than conventional CT scans. Measured by the Chi2-test.
One-year survival after randomization | 1 year
  To examine if MRI scans improves survival of patients with pancreatic cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Viborg Mortensen, Prof., Principal Investigator — Professor MTK AUh

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT05253313/Prot_SAP_000.pdf